CLINICAL TRIAL: NCT04433988
Title: Efficacy of Pentoxifylline as Add on Therapy in COVID19 Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional problems
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC-6-2020
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: COVID
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): 100 patients will receive standard treatment plus placebo
  Interventions: Drug: Placebo
- Pentoxifylline group (Experimental): 100 patients will receive standard treatment plus pentoxifylline 1200 mg/day
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400 mg SR tablet
  Arms: Pentoxifylline group
Drug: Placebo — Placebo tablet
  Arms: Control group

SUMMARY:
With potential antiviral effects on severe acute respiratory syndrome (SARS) and as a methyl-xanthine derived inhibitor of phosphodiesterase-4, pentoxifylline basically functions as a hemorrheologic agent for a better circulation and oxygenation and exerts unique effects on immune modulation, inflammation and oxidative stress. As the main regulator of cAMP metabolism, posphodiesterase-4 plays a key role in proinflammatory and immune cells. Pentoxifylline plays its anti-inflammatory role by reducing the production of proinflammatory cytokines such as TNF-a, IL-1 and IL-6. Given its unique impacts on immune modulation, homeostasis and fibrinolysis and its supportive effects on oxidative stress and organ failure, pentoxifylline can constitute a multipurpose and generally-safe adjuvant therapy for COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19 test
* Age >/= 18 y.o.

Exclusion Criteria:

* Allergic reaction to Pentoxifylline
* Ongoing anticoagulation
* History of GI bleeding
* History of Seizures
* Cardiac or other vascular stents
* History of severe renal disease
* History of intracranial hemorrhage.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-13 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 7 days
  Number of Participants need hospitalization

SECONDARY OUTCOMES:
Respiratory infection | 7 days
  Incidence of any acute respiratory infection
Serious Adverse Events | 7 days
  Absolute and relative frequencies of Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF